CLINICAL TRIAL: NCT05930210
Title: A Randomized, Double-Blind, Vehicle-controlled, Parallel, Phase III Study to Evaluate Efficacy and Safety of ENERGI-F703 GEL in Subjects With Diabetic Foot Ulcers
Brief Title: A Study to Evaluate ENERGI-F703 GEL in Diabetic Foot Ulcer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Energenesis Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENERGI-F703-04
Record Dates: First submitted 2023-06-15; First posted 2023-07-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Foot Ulcer; Foot Ulcer; Diabetes Mellitus; Wound
Keywords: Diabetic Foot Ulcer; Diabetes Mellitus; Wound Healing
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Diabetes Mellitus; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ENERGI-F703 GEL (Experimental): ENERGI-F703, topical application, 2 times daily for 16 weeks
  Interventions: Drug: ENERGI-F703 GEL
- ENERGI-F703 matched vehicle (Placebo Comparator): ENERGI-F703 matched vehicle, topical application, 2 times daily for 16 weeks
  Interventions: Drug: ENERGI-F703 matched vehicle

INTERVENTIONS:
Drug: ENERGI-F703 GEL — Standard of care and ENERGI-F703 GEL are applied for the treatment of diabetic foot ulcers.
  Arms: ENERGI-F703 GEL
Drug: ENERGI-F703 matched vehicle — Standard of care and ENERGI-F703 matched vehicle are applied for treatment of diabetic foot ulcers.
  Arms: ENERGI-F703 matched vehicle

SUMMARY:
This Phase 3 study is a randomized, double-blind, vehicle-controlled, multiple-center, parallel study to evaluate efficacy and safety of ENERGI-F703 GEL compared with vehicle control in subjects with Wagner Grade 1 to Grade 2 diabetic foot ulcers. Baseline target ulcer size (<16 cm2 vs ≥16 cm2 ) will be included as a stratification factor. Subjects will be randomized 1:1 to receive ENERGI-F703 GEL or vehicle control using an interactive web response system for randomization to automatically assign a unique subject randomization number. Total duration of the study will be up to 31 weeks including Screening visit (approximately 2 to 3 weeks), double-blind dosing/observation phase (16 weeks), and a safety follow-up of 12 weeks after the last administration of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years old.
2. Subject must have diagnosed with diabetes mellitus (DM), eg, currently under DM medication treatment or subjects with naïve DM with duplicated hemoglobin A1c over 6.5% and fasting plasma glucose over 126 mg/dL measured at least 1 week apart before screening.
3. Subject must have at least 1 cutaneous ulcer on the foot and not healing for at least 4 weeks. The largest diabetic foot ulcer will be selected as target ulcer. If 2 or more ulcers have the largest size, the one with worst grade will be selected. If 2 or more ulcers have the largest size and grade, the one with longest duration will be selected.
4. The target ulcer is classified as Grade 1 to Grade 2 ulcer according to Wagner Grading System and with ulcer size of 1.5 cm2 to 25 cm2.
5. Diabetic foot ulcers should be free of any necrosis or infection
6. Subject has signed the written informed consent form
7. Male subjects must be surgically sterile or commit to the use of a reliable method of birth control (must agree to use double-barrier contraception in the event of sexual activity) or be practicing abstinence for the duration of the study and for 30 days after study treatment administration.
8. Female subjects are eligible only if all of the following apply:

   * Not pregnant with a negative serum pregnancy test at Screening visit and negative urine pregnancy test within 24 hours before randomization (test not required for females of non-childbearing potential, defined as surgically sterile [eg, hysterectomy or bilateral oophorectomy] or postmenopausal [amenorrheic for at least 1 year])
   * Not lactating
   * Not planning to become pregnant during the study
   * If of childbearing potential, commits to the use of a highly effective method of contraception for the duration of the study and at least 30 days after study treatment administration.

Exclusion Criteria:

1. History or evidence of osteomyelitis as confirmed by the investigator. An x-ray/pathology assessment of debridement or a probe-to-bone (PTB) test will be used to determine presence of osteomyelitis. However, participants who have a history or evidence of osteomyelitis in other parts of their body are eligible to participate in the study. If the medical history of osteomyelitis was cured by antibiotic therapy, surgery or amputation for more than 1 year, and no recurrence, no finding to the current leg and foot after testing, the participant can be enrolled
2. With target ulcer size decreased by at least 30% after at least 2 weeks of standard of care-only period between screening and randomization
3. Subjects with highly exudated wounds which require dressing changes more than 3 times a day may be enrolled, but heavily exudated wounds should not be selected as target ulcers
4. With poor nutritional status (serum albumin <2g/dL or prealbumin <10 mg/dL), poor diabetic control (hemoglobin A1c >12%), a leukocyte counts <2,000/mm3, abnormal liver function (aspartate aminotransferase, alanine aminotransferase >3 x upper limit of normal range) within 21 days before Randomization visit
5. Requiring treatment with systemic corticosteroids, immunosuppressive or chemotherapeutic agents
6. With known or suspected hypersensitivity to any ingredients of study product and vehicle
7. With coronary heart disease with myocardial infarction, coronary artery bypass graft, or percutaneous transluminal coronary angioplasty within 3 months prior to study (patients who have undergone peripheral angioplasty should be excluded unless the surgery was performed at least 30 days prior to screening)
8. Known or suspected history of drug abuse or a recent history of alcohol abuse (regularly drinks >4 units of alcohol per day: 1 unit = 8 oz. beer, 3 oz. wine, or 1 oz. spirits) within 6 months prior to screening (within 6 months prior to screening includes both drug abuse and alcohol abuse)
9. History or positive test results for HIV
10. Malignancy in the last 2 years, with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix
11. Ankle brachial index <0.8 or >1.4
12. Enrollment in any investigational drug trial within 4 weeks before entering this study
13. With any condition judged by the investigator that entering the trial may be detrimental to the subject -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The ulcer complete closure rate | Weeks 16
  Proportion of subjects with a recording of complete ulcer closure at Week 16 (the end of the treatment period) as assessed by the investigator, where such closure is subsequently confirmed at 2 consecutive study visits over a 2-week period (ie, by Week 18). A complete ulcer closure is defined as 100% skin re epithelialization without drainage or dressing requirements.

SECONDARY OUTCOMES:
The time to ulcer closure | Weeks 4, 6, 8, 10, 12, 14, and 16
  Time to ulcer closure in weeks, defined as the time from randomization to first record of complete closure, as assessed by the investigator, where complete closure is subsequently confirmed at 2 consecutive study visits over a 2-week period
The frequency and severity of adverse events | Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, and 28
  Frequency and severity of adverse events (AEs), including treatment emergent AEs, serious AEs, treatment-related AEs, and treatment-related serious AEs
The proportion of subjects with complete ulcer closure | Weeks 4, 6, 8, 10, 12, 14, and 16
  Proportion of subjects with confirmed complete ulcer closure as assessed by the investigator.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (10):
  - A and D Doctor Center, Miami, Florida
  - Bioclinical Research, Miami, Florida
  - Reliant Medical Research, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - New Horizons Research, Palmetto Bay, Florida
  - IACT Health, Columbus, Georgia
  - The Jackson Clinic PA, Jackson, Tennessee
  - Mt. Olympus Medical Research, Houston, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Salem Veterans Affairs Medical Center VAMC, Salem, Virginia
- Taiwan (14):
  - Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Kung Tien General Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Cathay General Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Shin Kong Wu Ho Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided